CLINICAL TRIAL: NCT00479843
Title: Development of a Programme to Show the Positive Effect of a Nutritional Programme on Preventing Functional and Weight Losses in Patients With Dementia
Brief Title: Nutritional Programme for Dementia Elderly Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Institut Català de l'envelliment, Barcelona, Spain (Unknown); Hospital Purpan (Other); NESTEC R&D, Switzerland (Unknown); Group MAPI-NAXIS, CRO, Lyon, France (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05.19.CLI
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer Disease; Dementia; Elderly; Nutrition; Malnutrition; Weight Loss
MeSH Terms: conditions — Alzheimer Disease; Dementia; Malnutrition; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Nutritional programme

SUMMARY:
The main objective of this study is the improvement of the quality of life and state of health of elderly people with cognitive deterioration and their families through a weight loss prevention programme.

The secondary objectives are the improvement of the state of nutrition, a reduction in the use of resources and a reduction in the burden on the main carer.

DETAILED DESCRIPTION:
Main objective The main objective of this project is the evaluation of the effectiveness of a nutrition programme in patients with Alzheimer's or other dementias. Through the Nutrition Programme the idea is to reduce functional and weight loss in elderly people with cognitive deterioration and their families.

Evaluation of the effectiveness of the intervention

-The main evaluation criteria which will allow the effectiveness of this intervention to be evaluated are the reduction in the loss of autonomy measured by the DA/IDA scale.

Secondary objectives

The secondary objectives of this study are:

* Improvement in the patient's state of nutrition The measurement criteria which will allow the patient's nutritional state to be evaluated will be their weight, BMI and MNA.
* Reducing the burden on carers. The Zarit scale will be used for this evaluation.
* Evaluation of the use of healthcare and social resources. The RUD scale will be used.
* Improvement of medical practice regarding nutrition.
* Evaluation of the representatives of our population with regard to the participation in a programme of these characteristics evaluating.
* Evaluation of the satisfaction of elderly people and their families in relation to the programme.

ELIGIBILITY:
Inclusion Criteria:

* The patient has dementia according to DSM IV criteria.
* The patient has an MMSE less than or equal to 26.
* The patient lives in his/her home.
* The patient is in the charge of a carer.
* Informed consent for participation in the study by the responsible relative and, if possible, from the patient or legal guardian.

Exclusion Criteria:

* The patient lives in an institution.
* The patient is in a terminal situation.
* The patient does not have a main carer.
* Patient has a nasogastric feed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of the intervention -The main evaluation criteria which will allow the effectiveness of this intervention to be evaluated are the reduction in the loss of autonomy measured by the DA/IDA scale. | Baseline, 6 months, 12 months

SECONDARY OUTCOMES:
-Improvement in the patient's state of nutrition -Reducing the burden on carers with the Zarit scale. -Evaluation of the use of healthcare and social resources with the RUD scale. -Improvement of medical practice regarding nutrition. | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoni SALVA, MD, Principal Investigator — SPAIN: Institut Català de l'envelliment
Locations (1):
- Institut Català de l'envelliment, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Salvà A(1) , Fernández E(2), Andrieux S(3), Schiffrin E(4), Vellas B(3), y el grupo Nutrialz. 1. Institut de l'Envelliment. Universitat Autònoma de Barcelona. 2. Service de Gerontologie Clinique. Hôpital Pourpan. Caselardit. Toulouse. France. 3. Nestle Nutrition. Vevey. Switzerland. Estado nutricional de un grupo de pacientes ambulatorios y las principales correlaciones con las variables de la valoración geriátrica: El Estudio Nutrialz.49th Congress from the spanish aging association (6-9 June 2007, Palma de Mallorca) Salvà A(1) , Fernández E(2), Andrieux S(3), Schiffrin E(4), Vellas B(3), y el grupo Nutrialz. 1. Institut de l'Envelliment. Universitat Autònoma de Barcelona. 2. Service de Gerontologie Clinique. Hôpital Pourpan. Caselardit. Toulouse. France. 3. Nestle Nutrition. Vevey. Switzerland Nutritional status for ambulatory dementia patients and its main correlation with caregivers psychosocial variables: The Nutrialz Study INTERNATIONAL ASSOCIATION OF GERONTOLOGY AND GERIATRICS VI EUROPEAN CONGRESS (5-8 July 2007, Saint Petersburg).
- [Derived] Roque M, Salva A, Vellas B. Malnutrition in community-dwelling adults with dementia (NutriAlz Trial). J Nutr Health Aging. 2013 Apr;17(4):295-9. doi: 10.1007/s12603-012-0401-9. PMID 23538648
- [Derived] Salva A, Roque M, Rojano X, Inzitari M, Andrieu S, Schiffrin EJ, Guigoz Y, Vellas B. Falls and risk factors for falls in community-dwelling adults with dementia (NutriAlz trial). Alzheimer Dis Assoc Disord. 2012 Jan-Mar;26(1):74-80. doi: 10.1097/WAD.0b013e318215ca90. PMID 22354139
- [Derived] Salva A, Andrieu S, Fernandez E, Schiffrin EJ, Moulin J, Decarli B, Rojano-i-Luque X, Guigoz Y, Vellas B; NutriAlz group. Health and nutrition promotion program for patients with dementia (NutriAlz): cluster randomized trial. J Nutr Health Aging. 2011 Dec;15(10):822-30. doi: 10.1007/s12603-011-0363-3. PMID 22159768